CLINICAL TRIAL: NCT06803797
Title: A Behavior Change Technique (BCT) Intervention to Develop a Walking Habit Among Caregivers for Persons With Alzheimer's Disease (AD) or Alzheimer's Disease Related Dementias (ADRD)
Brief Title: BCT Intervention For Walking Habit Among Caregivers of People With AD/ADRD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 24-0045; 2P30AG063786 (NIH)
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Inactivity, Physical
Keywords: caregiver; Alzheimer's disease; Alzheimer Related Dementia; physical activity; behavior change techniques; habit formation
MeSH Terms: conditions — Sedentary Behavior; Alzheimer Disease; Motor Activity

STUDY DESIGN:
Intervention Model Description: This will be a 12-week, NIH Stage II Behavioral Trial, consisting of a single-arm, multi-component, personalized BCT intervention trial, enrolling caregivers of persons with AD/ADRD. Participants will be provided with 4 BCTs daily (Goal Setting, Action Planning, Self-Monitoring, and Prompt/Cue) that have been associated with habit formation theory and development of physical activity habits in prior research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): This will be a 12-week, single-arm, multi-component, personalized BCT intervention. We will provide participants with 4 BCTs daily (Goal Setting, Action Planning, Self-Monitoring, and Prompt/Cue) that have been associated with habit formation theory and development of physical activity habits in prior research.
  Interventions: Behavioral: Behavior Change Technique Package

INTERVENTIONS:
Behavioral: Behavior Change Technique Package — Behavior Change Technique 1: Goal setting (Behavior) (BCT 1.1). Goal setting for behavior is defined as setting a goal for the behavior to be achieved.
  Behavior Change Technique 2: Action planning (BCT 1.4). Action planning is defined as detailing the plan of where, for how long, and at what time taking medication is going to be performed.
  Behavior Change Technique 3: Self-monitoring of behavior (BCT 2.3). Self-monitoring of behavior is defined as monitoring and recording behavior.
  Behavior Change Technique 4: Prompts/Cues (BCT 7.1) This BCT is defined as prompt rehearsal and repetition of the behavior in the same context repeatedly, so that the context elicits the behavior.

SUMMARY:
This 12-week trial will test the efficacy of a multi-component, personalized text-message delivered behavior change technique (BCT) intervention to encourage habitual physical activity (defined as regular walking of 1,000 or more steps during a one-hour period on 7 consecutive days according to a personalized walking plan) among care providers of persons with AD/ADRD via the key mechanism of behavior change (MoBC) of automaticity.

The main question it aims to answer whether a multi-component, personalized BCT intervention to increase a walking habit of 1,000 steps/day will lead to successful development of habitual walking among 60 percent of caregivers enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Identify as a caregiver (formal/paid or informal/unpaid) for persons with Alzheimer's Disease or Alzheimer's Disease Related Dementias (AD/ADRD)
* Age >=18 and <=85
* Speak English or Spanish as primary language
* Self-report low levels of physical activity or walking

Exclusion Criteria:

* Individuals who self-report having been informed by a clinician it is medically or physically unsafe to engage in a walking intervention
* Does not own or cannot regularly access a smartphone capable of receiving text messages or accessing the internet
* Does not own or have access to an email address
* Lives outside the United States

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Binary indicator of habit formation | Baseline to intervention period (12 weeks)
  Binary indicator of habit formation, defined as a daily walking habit of 1,000 steps during a pre-determined period identified during baseline. Assessing the efficacy of the personalized BCT intervention by testing the null hypothesis of habit formation rate equal to 40% using a 1-sample binomial test at the 5% level 2-sided. Rate of habit formation will be summarized using the observed proportion, along with a 95% confidence interval.

SECONDARY OUTCOMES:
Habit formation association with changes in automaticity | Baseline (first 2 weeks of study) and last 2 weeks of intervention
  Examine whether habit formation will be associated with positive changes in automaticity, using Fisher's exact test (5% 2-sided). Specifically, for each participant, the difference between average automaticity during the last 2 weeks of intervention and average baseline automaticity will be calculated. Rate of habit formation between the group of participants, whose automaticity increased and the participants whose automaticity did not, will be compared using a Fisher's exact test. Logistic regression will be used to assess the effects of automaticity on the development of a daily walking habit with adjustment for other factors, such caregiver demographic characteristics and factors related to caregiving.
Longitudinal association between automaticity and habitual walking over time | Baseline to intervention period (12 weeks)
  Weekly automaticity and its association with habit formation using a multivariate Bayesian logistic regression model, trained using iPIPE,238 a novel statistical learning method.
Heterogeneity of treatment effects for habit formation and on changes in automaticity | Baseline to intervention period (12 weeks)
  Conduct analyses of heterogeneity of treatment effects (HTEs) across participants. This will involve examining the heterogeneity in time to achieving habitual daily walking due to the BCT intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Butler, PhD, Principal Investigator — Northwell Health
Locations (1):
- Institute of Health System Science, New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Scientific data generated as a result of this research will be shared broadly via OpenScience: https://cos.io/ or a comparable data registry. There will be no identifiable data posted publicly.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The study protocol, including the statistical analysis plan, will be made available in addition to the informed consent form following completion of recruitment but prior to publication of any data from the current study. De-identified individual participant data will be made available at time of primary outcome manuscript publication, whichever comes last. We anticipate this data to be available on the Open Science Framework or comparable data registry indefinitely.
Access Criteria: All de-identified study data and supporting information will be stored on the Open Science Framework or comparable data registry, a free web application with no access restrictions.

REFERENCES:
- [Derived] Miller D, Jordan L, Lambert S, Goodwin AM, Sinvani L, Perrin A, Cheung YK, Davidson KW, Butler MJ. Protocol for a single-arm, multi-component behavior change technique (BCT) intervention to develop a walking habit among caregivers for persons with Alzheimer's disease and related dementias (ADRD). Contemp Clin Trials. 2026 Jan 30:108248. doi: 10.1016/j.cct.2026.108248. Online ahead of print. PMID 41621469